CLINICAL TRIAL: NCT03763513
Title: Investigation of Acute Effect of Extracorporeal Shock Wave Therapy and Extracorporeal Shock Wave Therapy+Kinesyotaping on Pain and Grip Strength in Patients/Athletes With Lateral Epicondylitis
Brief Title: Investigation of Acute Effect of ESWT and ESWT+KT on Pain and Grip Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bihter Aslanyurek, Reserach Assistant. PhD. PT. Bihter Akınoğlu, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYBU
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain; Muscle Strength; Lateral Epicondylitis; Kinesio Taping
Keywords: Tennis Elbow; Taping; Grip Strength; Pain
MeSH Terms: conditions — Pain; Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Active Comparator): the first group:The group that will receive Extra corporeal shock wave therapy
  Interventions: Device: ESWT
- ESWT+KT (Experimental): the second group:The group that will receive Extra corporeal shock wave therapy + Kinesiotaping application
  Interventions: Device: ESWT; Other: Kinesiotaping Application

INTERVENTIONS:
Device: ESWT — Extracorporeal Shock Wave Therapy=ESWT
Other: Kinesiotaping Application — Kinesiotaping=KT (CT)
  Arms: ESWT+KT

SUMMARY:
The aim of this study was to investigate the acute effect of CT application in combination with ESWT and ESWT on pain and grip strength in athletes/patients with lateral epicondylitis.It is planned that at least 30 athletes aged 18-40 who are at the Ministry of Youth and Sports, Ministry of Health, Ministry of Health Affairs and who have been diagnosed with LE by specialist doctor.

After taking the information about birth dates, height, weight and dominant sides of the athletes who are willing to participate in the study, pain intensities and hand grip strengths will be evaluated. Then the athletes will be randomly divided into 2 groups according to closed envelope method. First group ESWT application; 4 sessions will be held for 4 weeks. The second group included ESWT + CT; 4 sessions will be held for 4 weeks. Pain severity and hand grip strength will be evaluated again after treatment.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE); the most common cause of elbow pain. It is typically characterized by pain around the lateral epicondyle during resistant wrist extension. This condition has been reported to occur as a result of degenerative angiofibroblastic hyperplasia of the wrist extensor tendons due to repetitive microtrauma. Although conservative treatments are usually used in lateral epicondylitis, many of them do not have sufficient evidence. In some cases, the healing phase lasts for months, which may be long enough to affect quality of life and sport performance.

Extracorporeal shock wave therapy (ESWT) is used in musculoskeletal problems with a possible mechanism of action, including hyperstimulation analgesia, neovascularization, and induction of the healing process. However, this method is a painful method due to the shock wave applied and may cause temporary redness in the area of application. This may cause the subcutaneous fascia of the affected area to be affected by the application pressure. Kinesiotaping (KT) is widely used in the treatment of various musculoskeletal problems. The band, invented by the Japanese chiropractor Kenzo Kase in the 1970s, is a heat-sensitive acrylic adhesive and an elastic woven cotton stripe with a maximum tensile strength of up to about 40-60% of its total length. Many effects of KT have been hypothesised, including improvement of feedback and correction of the articular alignment disorder. KT has an effect on the skin and fascia. recovery will be provided faster.

The aim of this study is to compare the effects of ESWT application with ESWT + KT application. In this study, our hypothesis is that ESWT + KT application will have more effect on pain and muscle strength in LE patients than ESWT alone.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Lateral Epicondylitis Disease
* has been doing professional sports for at least three years

Exclusion Criteria:

* Having systemic problems,
* Having health problems,
* Has undergone any surgical operation in the upper extremity
* Has suffered upper extremity injury in the last three months
* Lack of inclusion criteria
* Neurological and orthopedic problems of the upper extremity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Level: visual analog scale | 4 weeks
  The pain level will evaluate By visual analog scale;min:0=no pain, maximum 10=irresistible pain
Muscle Strength | 4 weeks
  The muscle strength will evaluate by hand grip strength by dynamometer, is evaluating by mmHg bigger means stronger

SECONDARY OUTCOMES:
Disability Level/Functionality | 4 weeks
  By the DASH (Disability arm shoulder hand) questionaire, min =0, maks 100 the bigger point means worse functionality